CLINICAL TRIAL: NCT02383472
Title: Transcranial LED Therapy for the Treatment of Chronic Mild Traumatic Brain Injury
Brief Title: LED Therapy for the Treatment of Concussive Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Football League (Other)
Responsible Party: Principal Investigator, William Meehan III, MD, Director of Research - Sports Medicine, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-P00002527
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Results first posted 2018-06-29 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-06

CONDITIONS: Brain Concussion
Keywords: Concussion; Mild Traumatic Brain Injury; MTBI; LED; Light Emitting Diode; Headache; Brain Concussion
MeSH Terms: conditions — Brain Concussion; Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MedX Health Console model 1100 (Experimental): The treatment group will receive LED treatments over 6 weeks, 3 times per week, totaling 18 visits. All treatments will take place at Boston Children's Hospital. The cluster heads are applied to frontal, parietal, and temporal areas. Each cluster head is applied to the forehead/scalp areas for up to 10 minutes. There will be two 10-minute LED/placebo treatment periods per visit, each with different cluster head placements on the head/scalp.
  Interventions: Device: MedX Health Console model 1100
- MedX Health Console model 1100-placebo (Placebo Comparator): Subjects enrolled in the placebo group will be on the same schedule as the treatment group. The placebo group will receive LED placebo over 6 weeks, 3 times per week, totaling 18 visits. All placebo patients will take place at Boston Children's Hospital. The cluster heads are applied to frontal, parietal, and temporal areas. Each cluster head is applied to the forehead/scalp areas for up to 10 minutes. There will be two 10-minute LED/placebo treatment periods per visit, each with different cluster head placements on the head/scalp.
  Interventions: Device: MedX Health Console model 1100-placebo

INTERVENTIONS:
Device: MedX Health Console model 1100 — All treatments will be administered using the MedX Health Console model 1100. These units were cleared by the FDA as non-significant risk in 2003 and approved for home treatment use in 2005 "for temporary increase in local blood flow circulation . . . for temporary relief of minor muscle and joint aches." Cluster heads are 2 inches in diameter. Each contains 9 red (633nm wavelength) diodes and 52 near infrared (870 nm wavelength) diodes. LED cluster heads would be applied to the frontal, parietal and temporal areas, as well as the mid sagittal suture line
  Other Names: MedX LCT 100 & Duolight; Manufacturer-MedX Health Inc.
  Arms: MedX Health Console model 1100
Device: MedX Health Console model 1100-placebo — The placebo machine is identical in appearance as the treatment machine; It vibrates, warms, and does everything the treatment machine does except it does not have LED lights on the marker, therefore it cannot emit light. Subjects enrolled in the placebo group will be on the same schedule as the treatment group. They will have two, 10 minute treatments, three times a week totaling 18 visits. The placebo allows the researchers to isolate the effect of the study treatment. If patient's in the LED treatment group fare significantly better than those in the placebo treatment group, the study helps support the conclusion that the LED therapy is effective.
  Other Names: MedX LCT 100 & Duolight; Manufacturer-MedX Health Inc.
  Arms: MedX Health Console model 1100-placebo

SUMMARY:
A double blind randomized trial of light-emitting diode (LED) therapy for patients suffering from mild traumatic brain injury (mTBI). Patients seen in the Sports Concussion Clinic with cognitive symptoms lasting for greater than 4 weeks will be randomized to either placebo therapy (controls) or treatment with LED therapy (cases). Both cases and controls would complete post-concussion symptom scales Delis-Kaplan Executive Function System (D-KEFS), and ImPACT studies on entry into the study and at weeks 3 and 6, or earlier if their symptoms resolve before the end of the 6 week period.

DETAILED DESCRIPTION:
Concussion, also known as mild traumatic brain injury (mTBI), results from a rotational acceleration of the brain. The biomechanical forces which cause concussion lead to the opening of ion channels within the neuronal cell membranes, allowing for a massive influx of sodium and efflux of potassium. This results in a spreading depression type of phenomenon, leading to the depolarization of neurons diffusely throughout the brain.19 In order to restore the homeostatic ion gradients across the membrane, the sodium-potassium pumps require increasing amounts of adenosine triphosphate (ATP). Thus, there is an increased need for ATP after concussion. ATP is supplied by the glycolysis of glucose from the blood stream. Both experimental models of concussion and human studies, however, show decreased cerebral blood flow after the initial response to injury. Thus, there is an increased demand for ATP after concussion; but a diminished supply of glucose to meet the demand.

The absorption of light in the red/near infrared wavelength spectrum by cytochrome C oxidase increases ATP synthesis. Thus, by increasing ATP synthesis, red/near infrared LEDs can treat the underlying pathophysiological cause of concussion symptoms. If successful, this would be the first therapy to directly treat the underlying pathophysiology of concussion.

ELIGIBILITY:
Inclusion Criteria:

* Patients 11 years old or greater
* Diagnosed with a concussion whose symptoms have persisted for more than 4 weeks
* Total score on the cognitive components of the post-concussion symptom scale exceeds 9, or if they have a composite score on any one of the 4 main outputs of the computerized neurocognitive assessment: Immediate Post-concussion Assessment and Cognitive Testing (ImPACT) that is below the 90th percentile for their age.

Exclusion Criteria:

* Clinically indicated imaging has been obtained where a hemorrhage is demonstrated
* Being considered for an alternate diagnosis (other than concussion)
* Have a pre-injury diagnosis of any of the following: depression, post-traumatic stress disorder, other psychiatric disorder
* Taking any of the following medications: amantadine, , amphetamine, atomoxetine

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P Meehan, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Boston Children's Hospital at Waltham, Waltham, Massachusetts

REFERENCES:
- [Background] Naeser MA, Zafonte R, Krengel MH, Martin PI, Frazier J, Hamblin MR, Knight JA, Meehan WP 3rd, Baker EH. Significant improvements in cognitive performance post-transcranial, red/near-infrared light-emitting diode treatments in chronic, mild traumatic brain injury: open-protocol study. J Neurotrauma. 2014 Jun 1;31(11):1008-17. doi: 10.1089/neu.2013.3244. Epub 2014 May 8. PMID 24568233
- [Background] Hoge CW, McGurk D, Thomas JL, Cox AL, Engel CC, Castro CA. Mild traumatic brain injury in U.S. Soldiers returning from Iraq. N Engl J Med. 2008 Jan 31;358(5):453-63. doi: 10.1056/NEJMoa072972. Epub 2008 Jan 30. PMID 18234750
- [Background] Cantu RC. Chronic traumatic encephalopathy in the National Football League. Neurosurgery. 2007 Aug;61(2):223-5. doi: 10.1227/01.NEU.0000255514.73967.90. No abstract available. PMID 17762733
- [Background] Collins MW, Lovell MR, Iverson GL, Cantu RC, Maroon JC, Field M. Cumulative effects of concussion in high school athletes. Neurosurgery. 2002 Nov;51(5):1175-9; discussion 1180-1. doi: 10.1097/00006123-200211000-00011. PMID 12383362
- [Background] Gronwall D, Wrightson P. Cumulative effect of concussion. Lancet. 1975 Nov 22;2(7943):995-7. doi: 10.1016/s0140-6736(75)90288-3. PMID 53547
- [Background] Guskiewicz KM, Marshall SW, Bailes J, McCrea M, Cantu RC, Randolph C, Jordan BD. Association between recurrent concussion and late-life cognitive impairment in retired professional football players. Neurosurgery. 2005 Oct;57(4):719-26; discussion 719-26. doi: 10.1093/neurosurgery/57.4.719. PMID 16239884
- [Background] Guskiewicz KM, Mihalik JP, Shankar V, Marshall SW, Crowell DH, Oliaro SM, Ciocca MF, Hooker DN. Measurement of head impacts in collegiate football players: relationship between head impact biomechanics and acute clinical outcome after concussion. Neurosurgery. 2007 Dec;61(6):1244-52; discussion 1252-3. doi: 10.1227/01.neu.0000306103.68635.1a. PMID 18162904
- [Background] Guskiewicz KM, McCrea M, Marshall SW, Cantu RC, Randolph C, Barr W, Onate JA, Kelly JP. Cumulative effects associated with recurrent concussion in collegiate football players: the NCAA Concussion Study. JAMA. 2003 Nov 19;290(19):2549-55. doi: 10.1001/jama.290.19.2549. PMID 14625331
- [Background] Jordan BD, Relkin NR, Ravdin LD, Jacobs AR, Bennett A, Gandy S. Apolipoprotein E epsilon4 associated with chronic traumatic brain injury in boxing. JAMA. 1997 Jul 9;278(2):136-40. PMID 9214529
- [Background] McKee AC, Cantu RC, Nowinski CJ, Hedley-Whyte ET, Gavett BE, Budson AE, Santini VE, Lee HS, Kubilus CA, Stern RA. Chronic traumatic encephalopathy in athletes: progressive tauopathy after repetitive head injury. J Neuropathol Exp Neurol. 2009 Jul;68(7):709-35. doi: 10.1097/NEN.0b013e3181a9d503. PMID 19535999
- [Background] Omalu BI, DeKosky ST, Hamilton RL, Minster RL, Kamboh MI, Shakir AM, Wecht CH. Chronic traumatic encephalopathy in a national football league player: part II. Neurosurgery. 2006 Nov;59(5):1086-92; discussion 1092-3. doi: 10.1227/01.NEU.0000245601.69451.27. PMID 17143242
- [Background] Beauchamp K, Mutlak H, Smith WR, Shohami E, Stahel PF. Pharmacology of traumatic brain injury: where is the "golden bullet"? Mol Med. 2008 Nov-Dec;14(11-12):731-40. doi: 10.2119/2008-00050.Beauchamp. Epub 2008 Aug 18. PMID 18769636
- [Background] Mittenberg W, Burton DB. A survey of treatments for post-concussion syndrome. Brain Inj. 1994 Jul;8(5):429-37. doi: 10.3109/02699059409150994. PMID 7951205
- [Background] Zafonte R, Friedewald WT, Lee SM, Levin B, Diaz-Arrastia R, Ansel B, Eisenberg H, Timmons SD, Temkin N, Novack T, Ricker J, Merchant R, Jallo J. The citicoline brain injury treatment (COBRIT) trial: design and methods. J Neurotrauma. 2009 Dec;26(12):2207-16. doi: 10.1089/neu.2009.1015. PMID 19803786
- [Background] Meehan WP 3rd. Medical therapies for concussion. Clin Sports Med. 2011 Jan;30(1):115-24, ix. doi: 10.1016/j.csm.2010.08.003. PMID 21074086
- [Background] Meehan WP 3rd, Bachur RG. Sport-related concussion. Pediatrics. 2009 Jan;123(1):114-23. doi: 10.1542/peds.2008-0309. PMID 19117869
- [Background] Ommaya AK, Gennarelli TA. Cerebral concussion and traumatic unconsciousness. Correlation of experimental and clinical observations of blunt head injuries. Brain. 1974 Dec;97(4):633-54. doi: 10.1093/brain/97.1.633. No abstract available. PMID 4215541
- [Background] Giza CC, Hovda DA. The Neurometabolic Cascade of Concussion. J Athl Train. 2001 Sep;36(3):228-235. PMID 12937489
- [Background] Yamakami I, McIntosh TK. Effects of traumatic brain injury on regional cerebral blood flow in rats as measured with radiolabeled microspheres. J Cereb Blood Flow Metab. 1989 Feb;9(1):117-24. doi: 10.1038/jcbfm.1989.16. PMID 2910893
- [Background] Yoshino A, Hovda DA, Kawamata T, Katayama Y, Becker DP. Dynamic changes in local cerebral glucose utilization following cerebral conclusion in rats: evidence of a hyper- and subsequent hypometabolic state. Brain Res. 1991 Oct 4;561(1):106-19. doi: 10.1016/0006-8993(91)90755-k. PMID 1797338
- [Background] Yuan XQ, Prough DS, Smith TL, Dewitt DS. The effects of traumatic brain injury on regional cerebral blood flow in rats. J Neurotrauma. 1988;5(4):289-301. doi: 10.1089/neu.1988.5.289. PMID 3249308
- [Background] Mochizuki-Oda N, Kataoka Y, Cui Y, Yamada H, Heya M, Awazu K. Effects of near-infra-red laser irradiation on adenosine triphosphate and adenosine diphosphate contents of rat brain tissue. Neurosci Lett. 2002 May 3;323(3):207-10. doi: 10.1016/s0304-3940(02)00159-3. PMID 11959421
- [Background] Yu W, Naim JO, McGowan M, Ippolito K, Lanzafame RJ. Photomodulation of oxidative metabolism and electron chain enzymes in rat liver mitochondria. Photochem Photobiol. 1997 Dec;66(6):866-71. doi: 10.1111/j.1751-1097.1997.tb03239.x. PMID 9421973
- [Background] Oron A, Oron U, Streeter J, de Taboada L, Alexandrovich A, Trembovler V, Shohami E. low-level laser therapy applied transcranially to mice following traumatic brain injury significantly reduces long-term neurological deficits. J Neurotrauma. 2007 Apr;24(4):651-6. doi: 10.1089/neu.2006.0198. PMID 17439348
- [Background] McCrory P, Meeuwisse W, Johnston K, Dvorak J, Aubry M, Molloy M, Cantu R. Consensus statement on concussion in sport - The 3rd international conference on concussion in sport held in Zurich, November 2008. PM R. 2009 May;1(5):406-20. doi: 10.1016/j.pmrj.2009.03.010. No abstract available. PMID 19627927
- [Background] Collins M, Lovell MR, Iverson GL, Ide T, Maroon J. Examining concussion rates and return to play in high school football players wearing newer helmet technology: a three-year prospective cohort study. Neurosurgery. 2006 Feb;58(2):275-86; discussion 275-86. doi: 10.1227/01.NEU.0000200441.92742.46. PMID 16462481
- [Background] Field M, Collins MW, Lovell MR, Maroon J. Does age play a role in recovery from sports-related concussion? A comparison of high school and collegiate athletes. J Pediatr. 2003 May;142(5):546-53. doi: 10.1067/mpd.2003.190. PMID 12756388
- [Background] Lovell MR, Collins MW, Iverson GL, Field M, Maroon JC, Cantu R, Podell K, Powell JW, Belza M, Fu FH. Recovery from mild concussion in high school athletes. J Neurosurg. 2003 Feb;98(2):296-301. doi: 10.3171/jns.2003.98.2.0296. PMID 12593614
- [Background] Lovell MR, Collins MW, Iverson GL, Johnston KM, Bradley JP. Grade 1 or "ding" concussions in high school athletes. Am J Sports Med. 2004 Jan-Feb;32(1):47-54. doi: 10.1177/0363546503260723. PMID 14754723
- [Background] Delis DC, Kramer JH, Kaplan E, Holdnack J. Reliability and validity of the Delis-Kaplan Executive Function System: an update. J Int Neuropsychol Soc. 2004 Mar;10(2):301-3. doi: 10.1017/S1355617704102191. No abstract available. PMID 15012851
- [Background] Stuss DT, Ely P, Hugenholtz H, Richard MT, LaRochelle S, Poirier CA, Bell I. Subtle neuropsychological deficits in patients with good recovery after closed head injury. Neurosurgery. 1985 Jul;17(1):41-7. doi: 10.1227/00006123-198507000-00007. PMID 4022286

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in the September of 2012 from the Concussion Clinic within the Department of Sports Medicine and lasted through the spring on 2016.
Groups:
- MedX Health Console Model 1100: The treatment group will receive LED treatments over 6 weeks, 3 times per week, totaling 18 visits. The cluster heads are applied to frontal, parietal, and temporal areas. Each cluster head is applied to the forehead/scalp areas for up to 10 minutes. There will be two 10-minute LED/placebo treatment periods per visit, each with different cluster head placements on the head/scalp.
  MedX Health Console model 1100: All treatments will be administered using the MedX Health Console model 1100. These units were cleared by the FDA as non-significant risk in 2003 and approved for home treatment use in 2005 "for temporary increase in local blood flow circulation . . . for temporary relief of minor muscle and joint aches." Cluster heads are 2 inches in diameter. Each contains 9 red (633nm wavelength) diodes and 52 near infrared (870 nm wavelength) diodes. LED cluster heads would be applied to the frontal, parietal and temporal areas, as well as the mid sagittal suture line
- MedX Health Console Model 1100-placebo: Subjects enrolled in the placebo group will be on the same schedule as the treatment group. The placebo group will receive LED placebo over 6 weeks, 3 times per week, totaling 18 visits. The cluster heads are applied to frontal, parietal, and temporal areas. Each cluster head is applied to the forehead/scalp areas for up to 10 minutes. There will be two 10-minute placebo treatment periods per visit, each with different cluster head placements on the head/scalp.
  MedX Health Console model 1100-placebo: The placebo machine is identical in appearance as the treatment machine; It vibrates, warms, and does everything the treatment machine does except it does not have LED lights on the marker, therefore it cannot emit light. The placebo allows the researchers to isolate the effect of the study treatment. If patient's in the LED treatment group fare significantly better than those in the placebo treatment group, the study helps support the conclusion that the LED therapy is effective.
Period: Overall Study
Arm/Group | MedX Health Console Model 1100 | MedX Health Console Model 1100-placebo
Started | 23 | 30
Completed | 22 | 29
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MedX Health Console Model 1100 | MedX Health Console Model 1100-placebo | Total
Number analyzed (Participants) | 22 | 29 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.55 (13.12) | 21.21 (13.25) | 21.35 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 32
  Male | 9 | 10 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 22 | 27 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Participants taking stimulant medications [Count of Participants; unit: Participants] | 10 | 14 | 24
Migraine Headache [Count of Participants; unit: Participants] | 2 | 7 | 9
Psychiatric hx [Count of Participants; unit: Participants]
  Undefined | 14 | 22 | 36
  Anxiety | 1 | 0 | 1
  Depression | 0 | 3 | 3
  PTSD | 1 | 0 | 1
Neurodevelopmental Diagnosis [Count of Participants; unit: Participants]
  ADHD | 5 | 2 | 7
  Learning Disability | 1 | 2 | 3
Prior Concussions [Mean (Full Range); unit: Concussions] | 3.5 [1 to 10] | 2 [1 to 6] | 2.5 [1 to 10]
Injury characteristics [Count of Participants; unit: Participants]
  Sport-related concussion | 14 | 22 | 36
  Loss of Consciousness | 3 | 3 | 6
  Amnesia | 8 | 10 | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Change in Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) Score at Baseline and 6 Weeks.
Description: The primary outcome is mean difference on composite scores of Immediate Post-Concussion Assessment and Cognitive Testing (ImPACT) between entry into the study and completion of treatment (visit 18, week 6) for both the LED group and the placebo group. The mean difference is calculated by taking the mean of differences of the entry scores minus the 6 week scores. There are 5 composite scores on the ImPACT test; verbal memory, visual memory, visual motor speed, reaction time, and symptom score. The ranges for these subscales are as follows: verbal memory and visual memory: 0-100, visual motor speed: 0-60, reaction time: 0-1.0, and symptom score: 0-132. A higher verbal memory, visual memory, and visual motor speed represent a better outcome, while a lower reaction time and lower symptom score represent a better outcome.
Time Frame: From baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- MedX Health Console Model 1100-placebo: Subjects enrolled in the placebo group will be on the same schedule as the treatment group. The placebo group will receive LED placebo over 6 weeks, 3 times per week, totaling 18 visits. The cluster heads are applied to frontal, parietal, and temporal areas. Each cluster head is applied to the forehead/scalp areas for up to 10 minutes. There will be two 10-minute LED/placebo treatment periods per visit, each with different cluster head placements on the head/scalp.
  MedX Health Console model 1100-placebo: The placebo machine is identical in appearance as the treatment machine except it does not have LED lights on the marker, therefore it cannot emit light. The placebo allows the researchers to isolate the effect of the study treatment. If patient's in the LED treatment group fare significantly better than those in the placebo treatment group, the study helps support the conclusion that the LED therapy is effective.
Arm/Group | MedX Health Console Model 1100 | MedX Health Console Model 1100-placebo
Number analyzed (Participants) | 22 | 29
Units on a scale
  Verbal Memory | -0.9 (17.11) | -5.78 (12.08)
  Visual Memory | 3.52 (14.82) | -7.26 (12.07)
  Visual Motor Speed | -2.04 (6.36) | -5.15 (5.04)
  Reaction Time | -0.001 (0.16) | 0.030 (0.18)
  Symptom Score | 10.14 (10.13) | 11.44 (19.07)

2. Secondary Outcome: Mean Difference in Change in Delis-Kaplan Executive Function System (D-KEF) Color-Word Interference and Trail Making Test Performance at Weeks 3 and 6.
Description: This measure indicates the mean differences in Delis-Kaplan Executive Function System (D-KEF) tests between entry into the study and 3 weeks and entry into the study and 6 weeks for both the LED group and the placebo group. The mean difference is calculated by taking the mean of differences of the entry scores minus the 3 week scores and the entry scores minus the 6 week scores. D-KEFs color-word interferences, made up of color naming, word reading, and inhibition, is measured in seconds, a smaller number represents a better outcome. Participants were given 90 seconds to complete color naming and word reading and 180 seconds to complete inhibition. D-KEFs trail making test, made up of number sequencing, letter sequencing, and number-letter sequencing, is measured in seconds, a faster speed (lower number) represents a better outcome. Participants were given 150 seconds to complete number and letter sequencing and 240 seconds to complete number-letter sequencing.
Time Frame: From baseline to 3 weeks and from baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- MedX Health Console Model 1100: The treatment group will receive LED treatments over 6 weeks, 3 times per week, totaling 18 visits. Treatments will take place at Boston Children's Hospital. The cluster heads are applied to frontal, parietal, and temporal areas. Each cluster head is applied to the forehead/scalp areas for up to 10 minutes. There will be two 10-minute LED/placebo treatment periods per visit, each with different cluster head placements on the head/scalp.
  MedX Health Console model 1100: All treatments will be administered using the MedX Health Console model 1100. These units were cleared by the FDA as non-significant risk in 2003 and approved for home treatment use in 2005 "for temporary increase in local blood flow circulation . . . for temporary relief of minor muscle and joint aches." Cluster heads are 2 inches in diameter. Each contains 9 red (633nm wavelength) diodes and 52 near infrared (870 nm wavelength) diodes. LED cluster heads would be applied to the frontal, parietal and temporal ar
- MedX Health Console Model 1100-placebo: Subjects enrolled in the placebo group will be on the same schedule as the treatment group. The placebo group will receive LED placebo over 6 weeks, 3 times per week, totaling 18 visits. Placebo patients will take place at Boston Children's Hospital. The cluster heads are applied to frontal, parietal, and temporal areas. Each cluster head is applied to the forehead/scalp areas for up to 10 minutes. There will be two 10-minute LED/placebo treatment periods per visit, each with different cluster head placements on the head/scalp.
  MedX Health Console model 1100-placebo: The placebo machine is identical in appearance as the treatment machine; It vibrates, warms, and does everything the treatment machine does except it does not have LED lights on the marker, therefore it cannot emit light. Subjects enrolled in the placebo group will be on the same schedule as the treatment group. They will have two, 10 minute treatments, three times a week totaling 18 visits. The placebo allows the r
Arm/Group | MedX Health Console Model 1100 | MedX Health Console Model 1100-placebo
Number analyzed (Participants) | 22 | 29
Seconds
  D-KEFs Color Naming - 3 Weeks | 3.27 (4.03) | 4.76 (8.88)
  D-KEFs Color Naming - 6 Weeks | 3.76 (5.12) | 4.07 (9.00)
  D-KEFs Word Reading - 3 Weeks | 0.95 (2.98) | 4.07 (10.05)
  D-KEFs Word Reading - 6 Weeks | 1.71 (3.73) | 3.44 (13.98)
  D-KEFs Inhibition - 3 Weeks | 7.64 (5.49) | 4.48 (17.00)
  D-KEFs Inhibition - 6 Weeks | 32.62 (9.13) | 31.59 (14.73)
  D-KEFs Number Sequencing - 3 weeks | -24.45 (15.04) | -21.17 (17.55)
  D-KEFs Letter Sequencing- 3 weeks | -28.41 (14.06) | -19.51 (20.15)
  D-KEFs Number-Letter Sequencing- 3 weeks | 8.00 (12.66) | 21.93 (32.19)
  D-KEFs Number Sequencing - 6 weeks | 11.33 (7.3) | 6.89 (10.78)
  D-KEFs Letter Sequencing- 6 weeks | 6.86 (4.29) | 10.59 (9.49)
  D-KEFs Number-Letter Sequencing- 6 weeks | 12.95 (13.28) | 19.81 (30.34)

3. Secondary Outcome: Mean Difference in Change in Delis-Kaplan Executive Function System (D-KEF) Verbal Fluency Performance at Weeks 3 and 6.
Description: This measure indicates the mean differences in Delis-Kaplan Executive Function System (D-KEF) tests between entry into the study and 3 weeks and entry into the study and 6 weeks for both the LED group and the placebo group. The mean difference is calculated by taking the mean of differences of the entry scores minus the 3 week scores and the entry scores minus the 6 week scores. D-KEFs Verbal Fluency Test, made up of letter fluency and category fluency, is measured by number of responses, a larger number represents a better outcome. Participants were given 60 seconds to complete each fluency test.
Time Frame: From baseline to 3 weeks and from baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | MedX Health Console Model 1100 | MedX Health Console Model 1100-placebo
Number analyzed (Participants) | 22 | 29
Correct responses
  D-KEFs Verbal Fluency- letters 3 weeks | -3.45 (6.52) | -6.10 (8.26)
  D-KEFs Verbal Fluency- letters 6 weeks | -6.71 (7.89) | -9.89 (11.34)
  D-KEFs Verbal Fluency- category 3 weeks | -1.14 (4.17) | -0.03 (4.12)
  D-KEFs Verbal Fluency- category 6 weeks | -1.62 (4.09) | -2.00 (4.62)

4. Secondary Outcome: Mean Difference in Change in Total Post Concussion Symptom Score (PCSS) at Weeks 3 and Weeks 6.
Description: This measure indicates the mean differences in total post concussion symptom score (PCSS) between entry into the study and 3 weeks and entry into the study and 6 weeks for both the LED group and the placebo group. The mean difference is calculated by taking the mean of differences of the entry scores minus the 3 week scores and the entry scores minus the 6 week scores. The PCSS is a sum of severity scores from 0-6 (0=none, 6=severe) for 22 individual symptoms, like headache, neck pain, or drowsiness. The range for the PCSS is 0-132, a lower score represents a better outcome.
Time Frame: From baseline to 3 weeks and from baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MedX Health Console Model 1100 | MedX Health Console Model 1100-placebo
Number analyzed (Participants) | 22 | 29
units on a scale
  PCSS Total Score - 3 Weeks | 9.41 (12.62) | 7.03 (16.96)
  PCSS Total score - 6 Weeks | 7.86 (14.5) | 14.63 (23.41)

5. Secondary Outcome: Mean Difference in Change in Total Cognitive Symptom Score at Weeks 3 and Weeks 6
Description: This measure indicates the mean difference in total cognitive symptom scores between entry into the study and 3 weeks and entry into the study and 6 weeks for both the LED group and the placebo group. The mean difference is calculated by taking the mean of differences of the entry scores minus the 3 week scores and the entry scores minus the 6 weeks scores. The total cognitive symptom scored is a sum of 7 symptom scores from the PCSS; feeling slowed down, feeling like "in a fog", "don't feel right", difficulty concentrating, difficulty remembering, fatigue or low energy, and confusion. The severity of these symptoms are scored 0-6, 0=none, 6=severe. The range for the total cognitive symptom score is 0-42, a lower score represents a better outcome.
Time Frame: From baseline to 3 weeks and from baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MedX Health Console Model 1100 | MedX Health Console Model 1100-placebo
Number analyzed (Participants) | 22 | 29
units on a scale
  Cognitive Sx Score - 3 Weeks | 3.95 (6.56) | 1.31 (6.96)
  Cognitive Sx Score - 6 Weeks | 4.00 (6.59) | 5.00 (8.95)

ADVERSE EVENTS:
Groups:
- MedX Health Console Model 1100: The treatment group will receive LED treatments over 6 weeks, 3 times per week, totaling 18 visits. All treatments will take place at Boston Children's Hospital. The cluster heads are applied to frontal, parietal, and temporal areas. Each cluster head is applied to the forehead/scalp areas for up to 10 minutes. There will be two 10-minute LED/placebo treatment periods per visit, each with different cluster head placements on the head/scalp.
  MedX Health Console model 1100: All treatments will be administered using the MedX Health Console model 1100. These units were cleared by the FDA as non-significant risk in 2003 and approved for home treatment use in 2005 "for temporary increase in local blood flow circulation . . . for temporary relief of minor muscle and joint aches." Cluster heads are 2 inches in diameter. Each contains 9 red (633nm wavelength) diodes and 52 near infrared (870 nm wavelength) diodes. LED cluster heads would be applied to the frontal, parietal and temporal ar
- MedX Health Console Model 1100-placebo: Subjects enrolled in the placebo group will be on the same schedule as the treatment group. The placebo group will receive LED placebo over 6 weeks, 3 times per week, totaling 18 visits. All placebo patients will take place at Boston Children's Hospital. The cluster heads are applied to frontal, parietal, and temporal areas. Each cluster head is applied to the forehead/scalp areas for up to 10 minutes. There will be two 10-minute LED/placebo treatment periods per visit, each with different cluster head placements on the head/scalp.
  MedX Health Console model 1100-placebo: The placebo machine is identical in appearance as the treatment machine; It vibrates, warms, and does everything the treatment machine does except it does not have LED lights on the marker, therefore it cannot emit light. Subjects enrolled in the placebo group will be on the same schedule as the treatment group. They will have two, 10 minute treatments, three times a week totaling 18 visits. The placebo allows the r
Arm/Group | MedX Health Console Model 1100 | MedX Health Console Model 1100-placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/30
Other Adverse Events (participants affected / at risk) | 1/23 | 0/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MedX Health Console Model 1100 (N=23) | MedX Health Console Model 1100-placebo (N=30)
Discomfort (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Patient complained cluster heads were "uncomfortable and hot"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No